CLINICAL TRIAL: NCT02296138
Title: A Randomised, Double-blind, Active-controlled Parallel Group Study to Evaluate the Effect of 52 Weeks of Once Daily Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination Compared With Tiotropium on Chronic Obstructive Pulmonary Disease (COPD) Exacerbation in Patients With Severe to Very Severe COPD. [DYNAGITO]
Brief Title: Comparing the Efficacy of Tiotropium + Olodaterol (5/5 µg) Fixed Dose Combination (FDC) Over Tiotropium 5µg in Reducing Moderate to Severe Exacerbations in Patients With Severe to Very Severe Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.19; 2014-002275-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-11-19; First posted 2014-11-20 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- tiotropium + olodaterol high dose (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: olodaterol; Drug: tiotropium
- tiotropium (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium

INTERVENTIONS:
Drug: olodaterol — fixed dose combination
  Arms: tiotropium + olodaterol high dose
Drug: tiotropium — fixed dose combination
  Arms: tiotropium + olodaterol high dose
Drug: tiotropium
  Arms: tiotropium

SUMMARY:
The overall objective is to assess the effect of once daily tiotropium + olodaterol fixed dose combination compared to 5 µg tiotropium (both delivered with the Respimat® inhaler) on moderate to severe COPD exacerbation in patients with severe to very severe COPD.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients, 40 years of age or older.
* Diagnosis of COPD with a documented post-bronchodilator Forced expiratory volume in one second (FEV1)< 60% of predicted normal and a post-bronchodilator FEV1/ forced vital capacity (FVC) <70% at Visit 1
* Documented history of at least one moderate to severe COPD exacerbation in the previous 12 months requiring treatment with systemic corticosteroids and/or antibiotics and/or related hospitalization.
* Symptomatically stable as defined by: no evidence of COPD exacerbation requiring use of either antibiotics and/or steroids 4 weeks prior to visit 1 and no evidence of change in their usual COPD medication 4 weeks prior to visit 1.
* Current or ex-smokers with a smoking history of more than 10 pack years.

Exclusion criteria:

* Significant disease other than COPD.
* Clinically relevant abnormal baseline haematology, blood chemistry or creatinine > x2 ULN will be excluded regardless of clinical condition. ( A repeat laboratory evaluation can be conducted if deemed necessary by the investigator.)
* Current documented diagnosis of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma
* A diagnosis of thyrotoxicosis
* A history of myocardial infarction within 6 months of screening visit.
* Life-threatening cardiac arrhythmia.
* Known active tuberculosis.
* Any malignancy unless free of disease for at least 5 years (patients with treated basal cell carcinoma or squamous cell skin cancers are allowed).
* A history of cystic fibrosis.
* Clinically relevant bronchiectasis.
* Patients with severe emphysema requiring endobronchial interventions within 6 months prior to screening
* A history of significant alcohol or drug abuse in the opinion of the investigator.
* Patients who have undergone thoracotomy with pulmonary resection
* Patients being treated with oral or patch ß-adrenergics.
* Patients being treated with oral corticosteroid medication at unstable doses
* Patients being treated with antibiotics for any reasons within 4 weeks of screening visit
* Patients being treated with PDE4 inhibitors within 3 months of screening visit
* Patients who have taken an investigational drug within one month or six half-lives
* Pregnant or nursing women.
* Women of childbearing potential not using a highly effective method of birth control.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7903 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (818):
- United States (117):
  - 1237.19.10039 Boehringer Ingelheim Investigational Site, Andalusia, Alabama
  - 1237.19.10009 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1237.19.10077 Boehringer Ingelheim Investigational Site, Florence, Alabama
  - 1237.19.10115 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1237.19.10069 Boehringer Ingelheim Investigational Site, Flagstaff, Arizona
  - 1237.19.10085 Boehringer Ingelheim Investigational Site, Peoria, Arizona
  - 1237.19.10110 Boehringer Ingelheim Investigational Site, Lincoln, California
  - 1237.19.10118 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1237.19.10074 Boehringer Ingelheim Investigational Site, Poway, California
  - 1237.19.10157 Boehringer Ingelheim Investigational Site, Lafayette, Colorado
  - 1237.19.10142 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1237.19.10133 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1237.19.10093 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1237.19.10029 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.19.10106 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.19.10020 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1237.19.10000 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1237.19.10135 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1237.19.10145 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 1237.19.10066 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1237.19.10032 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1237.19.10080 Boehringer Ingelheim Investigational Site, Duluth, Georgia
  - 1237.19.10011 Boehringer Ingelheim Investigational Site, Gainesville, Georgia
  - 1237.19.10112 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 1237.19.10037 Boehringer Ingelheim Investigational Site, Eagle, Idaho
  - 1237.19.10130 Boehringer Ingelheim Investigational Site, O'Fallon, Illinois
  - 1237.19.10065 Boehringer Ingelheim Investigational Site, River Forest, Illinois
  - 1237.19.10122 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 1237.19.10063 Boehringer Ingelheim Investigational Site, Topeka, Kansas
  - 1237.19.10048 Boehringer Ingelheim Investigational Site, Bowling Green, Kentucky
  - 1237.19.10108 Boehringer Ingelheim Investigational Site, Fort Mitchell, Kentucky
  - 1237.19.10109 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1237.19.10095 Boehringer Ingelheim Investigational Site, Opelousas, Louisiana
  - 1237.19.10113 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1237.19.10139 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1237.19.10117 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1237.19.10083 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1237.19.10072 Boehringer Ingelheim Investigational Site, Hollywood, Maryland
  - 1237.19.10027 Boehringer Ingelheim Investigational Site, Fall River, Massachusetts
  - 1237.19.10138 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1237.19.10103 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 1237.19.10075 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1237.19.10034 Boehringer Ingelheim Investigational Site, Farmington Hills, Michigan
  - 1237.19.10082 Boehringer Ingelheim Investigational Site, Traverse City, Michigan
  - 1237.19.10043 Boehringer Ingelheim Investigational Site, Fridley, Minnesota
  - 1237.19.10096 Boehringer Ingelheim Investigational Site, Rochester, Minnesota
  - 1237.19.10031 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 1237.19.10101 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 1237.19.10051 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1237.19.10084 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1237.19.10097 Boehringer Ingelheim Investigational Site, Missoula, Montana
  - 1237.19.10060 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 1237.19.10081 Boehringer Ingelheim Investigational Site, Marlton, New Jersey
  - 1237.19.10094 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1237.19.10137 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 1237.19.10143 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 1237.19.10035 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1237.19.10014 Boehringer Ingelheim Investigational Site, Calabash, North Carolina
  - 1237.19.10098 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1237.19.10131 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1237.19.10049 Boehringer Ingelheim Investigational Site, Elizabeth City, North Carolina
  - 1237.19.10154 Boehringer Ingelheim Investigational Site, Gastonia, North Carolina
  - 1237.19.10104 Boehringer Ingelheim Investigational Site, Hickory, North Carolina
  - 1237.19.10087 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 1237.19.10053 Boehringer Ingelheim Investigational Site, Shelby, North Carolina
  - 1237.19.10062 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 1237.19.10008 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1237.19.10042 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1237.19.10127 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1237.19.10121 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1237.19.10148 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1237.19.10005 Boehringer Ingelheim Investigational Site, Delaware, Ohio
  - 1237.19.10147 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1237.19.10055 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1237.19.10146 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1237.19.10021 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1237.19.10129 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 1237.19.10140 Boehringer Ingelheim Investigational Site, Oaks, Pennsylvania
  - 1237.19.10003 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1237.19.10019 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1237.19.10006 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1237.19.10136 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1237.19.10151 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1237.19.10041 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1237.19.10126 Boehringer Ingelheim Investigational Site, Johnston, Rhode Island
  - 1237.19.10054 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1237.19.10086 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1237.19.10058 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1237.19.10023 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 1237.19.10030 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 1237.19.10024 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.19.10128 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.19.10144 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1237.19.10071 Boehringer Ingelheim Investigational Site, Myrtle Beach, South Carolina
  - 1237.19.10099 Boehringer Ingelheim Investigational Site, Old Point Station, South Carolina
  - 1237.19.10025 Boehringer Ingelheim Investigational Site, Rock Hill, South Carolina
  - 1237.19.10033 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.19.10036 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.19.10010 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1237.19.10007 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 1237.19.10070 Boehringer Ingelheim Investigational Site, Boerne, Texas
  - 1237.19.10107 Boehringer Ingelheim Investigational Site, Corsicana, Texas
  - 1237.19.10153 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1237.19.10047 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1237.19.10111 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1237.19.10059 Boehringer Ingelheim Investigational Site, Kingwood, Texas
  - 1237.19.10061 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1237.19.10050 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1237.19.10091 Boehringer Ingelheim Investigational Site, Abingdon, Virginia
  - 1237.19.10076 Boehringer Ingelheim Investigational Site, Lynchburg, Virginia
  - 1237.19.10040 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1237.19.10089 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1237.19.10123 Boehringer Ingelheim Investigational Site, Everett, Washington
  - 1237.19.10120 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1237.19.10092 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1237.19.10001 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
  - 1237.19.10016 Boehringer Ingelheim Investigational Site, West Allis, Wisconsin
- Argentina (17):
  - 1237.19.54015 Boehringer Ingelheim Investigational Site, Bahía Blanca
  - 1237.19.54014 Boehringer Ingelheim Investigational Site, Berazategui
  - 1237.19.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1237.19.54004 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1237.19.54007 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1237.19.54011 Boehringer Ingelheim Investigational Site, Ciudad de Buenos Aires
  - 1237.19.54018 Boehringer Ingelheim Investigational Site, Ciudad de Buenos Aires
  - 1237.19.54010 Boehringer Ingelheim Investigational Site, La Plata
  - 1237.19.54012 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1237.19.54017 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1237.19.54019 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1237.19.54005 Boehringer Ingelheim Investigational Site, Mendoza
  - 1237.19.54006 Boehringer Ingelheim Investigational Site, Quilmes
  - 1237.19.54013 Boehringer Ingelheim Investigational Site, Rosario
  - 1237.19.54016 Boehringer Ingelheim Investigational Site, San Isidro
  - 1237.19.54001 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
  - 1237.19.54002 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- Australia (12):
  - 1237.19.61012 Boehringer Ingelheim Investigational Site, Campbelltown, New South Wales
  - 1237.19.61011 Boehringer Ingelheim Investigational Site, Kogarah, New South Wales
  - 1237.19.61008 Boehringer Ingelheim Investigational Site, Randwick, New South Wales
  - 1237.19.61010 Boehringer Ingelheim Investigational Site, Cairns, Queensland
  - 1237.19.61006 Boehringer Ingelheim Investigational Site, Chermside, Queensland
  - 1237.19.61001 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 1237.19.61002 Boehringer Ingelheim Investigational Site, Kent Town, South Australia
  - 1237.19.61007 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 1237.19.61013 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1237.19.61003 Boehringer Ingelheim Investigational Site, Melbourne, Victoria
  - 1237.19.61009 Boehringer Ingelheim Investigational Site, Parkville, Victoria
  - 1237.19.61004 Boehringer Ingelheim Investigational Site, Murdoch, Western Australia
- Austria (7):
  - 1237.19.43006 Boehringer Ingelheim Investigational Site, Feldbach
  - 1237.19.43004 Boehringer Ingelheim Investigational Site, Graz
  - 1237.19.43003 Boehringer Ingelheim Investigational Site, Leoben
  - 1237.19.43001 Boehringer Ingelheim Investigational Site, Linz
  - 1237.19.70001 Boehringer Ingelheim Investigational Site, Ryazan
  - 1237.19.43005 Boehringer Ingelheim Investigational Site, Salzburg
  - 1237.19.43002 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (7):
  - 1237.19.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.19.32007 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.19.32006 Boehringer Ingelheim Investigational Site, Gilly
  - 1237.19.32004 Boehringer Ingelheim Investigational Site, Jambes
  - 1237.19.32003 Boehringer Ingelheim Investigational Site, Lebbeke
  - 1237.19.32002 Boehringer Ingelheim Investigational Site, Turnhout
  - 1237.19.32005 Boehringer Ingelheim Investigational Site, Zichem
- Brazil (12):
  - 1237.19.55007 Boehringer Ingelheim Investigational Site, Belo Horizonte
  - 1237.19.55013 Boehringer Ingelheim Investigational Site, Botucatu
  - 1237.19.55011 Boehringer Ingelheim Investigational Site, Goiânia
  - 1237.19.55002 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.19.55006 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.19.55010 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.19.55012 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.19.55014 Boehringer Ingelheim Investigational Site, Santo André
  - 1237.19.55001 Boehringer Ingelheim Investigational Site, São Paulo
  - 1237.19.55005 Boehringer Ingelheim Investigational Site, São Paulo
  - 1237.19.55008 Boehringer Ingelheim Investigational Site, São Paulo
  - 1237.19.55009 Boehringer Ingelheim Investigational Site, Vitória
- Bulgaria (8):
  - 1237.19.35905 Boehringer Ingelheim Investigational Site, Plovdiv
  - 1237.19.35902 Boehringer Ingelheim Investigational Site, Rousse
  - 1237.19.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 1237.19.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 1237.19.35906 Boehringer Ingelheim Investigational Site, Sofia
  - 1237.19.35907 Boehringer Ingelheim Investigational Site, Troyan Municipality
  - 1237.19.35901 Boehringer Ingelheim Investigational Site, Varna
  - 1237.19.35908 Boehringer Ingelheim Investigational Site, Vidin
- Canada (38):
  - 1237.19.20011 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1237.19.20020 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1237.19.20016 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1237.19.20025 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1237.19.20035 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1237.19.20034 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 1237.19.20041 Boehringer Ingelheim Investigational Site, Maple Ridge, British Columbia
  - 1237.19.20010 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1237.19.20033 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1237.19.20036 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1237.19.20015 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1237.19.20021 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1237.19.20006 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 1237.19.20013 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1237.19.20018 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1237.19.20029 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1237.19.20009 Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - 1237.19.20019 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1237.19.20017 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1237.19.20026 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1237.19.20038 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1237.19.20022 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1237.19.20040 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1237.19.20030 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1237.19.20005 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.19.20037 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.19.20012 Boehringer Ingelheim Investigational Site, Waterloo, Ontario
  - 1237.19.20007 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 1237.19.20004 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 1237.19.20032 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1237.19.20008 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 1237.19.20014 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1237.19.20031 Boehringer Ingelheim Investigational Site, Saint-Charles-Borromée, Quebec
  - 1237.19.20023 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
  - 1237.19.20039 Boehringer Ingelheim Investigational Site, Trois-Rivières, Quebec
  - 1237.19.20003 Boehringer Ingelheim Investigational Site, Victoriaville, Quebec
  - 1237.19.20002 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - 1237.19.20027 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Chile (3):
  - 1237.19.53004 Boehringer Ingelheim Investigational Site, Quillota
  - 1237.19.53003 Boehringer Ingelheim Investigational Site, San Miguel
  - 1237.19.53002 Boehringer Ingelheim Investigational Site, Santiago
- Colombia (5):
  - 1237.19.57002 Boehringer Ingelheim Investigational Site, Bogotá
  - 1237.19.57004 Boehringer Ingelheim Investigational Site, Bogotá
  - 1237.19.57005 Boehringer Ingelheim Investigational Site, Bogotá
  - 1237.19.57003 Boehringer Ingelheim Investigational Site, Cali
  - 1237.19.57006 Boehringer Ingelheim Investigational Site, Medellín
- Croatia (3):
  - 1237.19.38501 Boehringer Ingelheim Investigational Site, Rijeka
  - 1237.19.38502 Boehringer Ingelheim Investigational Site, Zagreb
  - 1237.19.38503 Boehringer Ingelheim Investigational Site, Zagreb
- Czechia (10):
  - 1237.19.42001 Boehringer Ingelheim Investigational Site, Beroun
  - 1237.19.42010 Boehringer Ingelheim Investigational Site, Český Krumlov
  - 1237.19.42004 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1237.19.42002 Boehringer Ingelheim Investigational Site, Jindřichův Hradec
  - 1237.19.42006 Boehringer Ingelheim Investigational Site, Krnov
  - 1237.19.42007 Boehringer Ingelheim Investigational Site, Liberec
  - 1237.19.42003 Boehringer Ingelheim Investigational Site, Mělník
  - 1237.19.42005 Boehringer Ingelheim Investigational Site, Prague
  - 1237.19.42008 Boehringer Ingelheim Investigational Site, Prague
  - 1237.19.42009 Boehringer Ingelheim Investigational Site, Varnsdorf
- Denmark (8):
  - 1237.19.45004 Boehringer Ingelheim Investigational Site, Aalborg
  - 1237.19.45007 Boehringer Ingelheim Investigational Site, Aarhus
  - 1237.19.45006 Boehringer Ingelheim Investigational Site, Holstebro
  - 1237.19.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1237.19.45005 Boehringer Ingelheim Investigational Site, Kolding
  - 1237.19.45001 Boehringer Ingelheim Investigational Site, Odense
  - 1237.19.45008 Boehringer Ingelheim Investigational Site, Roskilde
  - 1237.19.45003 Boehringer Ingelheim Investigational Site, Vaerløse
- Finland (4):
  - 1237.19.35804 Boehringer Ingelheim Investigational Site, Helsinki
  - 1237.19.35805 Boehringer Ingelheim Investigational Site, Oulu
  - 1237.19.35801 Boehringer Ingelheim Investigational Site, Turku
  - 1237.19.35803 Boehringer Ingelheim Investigational Site, Turku
- France (19):
  - 1237.19.33016 Boehringer Ingelheim Investigational Site, Cannes
  - 1237.19.33014 Boehringer Ingelheim Investigational Site, La Tronche
  - 1237.19.33013 Boehringer Ingelheim Investigational Site, Marseille
  - 1237.19.33020 Boehringer Ingelheim Investigational Site, Marseille
  - 1237.19.33003 Boehringer Ingelheim Investigational Site, Montpellier
  - 1237.19.33024 Boehringer Ingelheim Investigational Site, Nantes
  - 1237.19.33017 Boehringer Ingelheim Investigational Site, Nice
  - 1237.19.33018 Boehringer Ingelheim Investigational Site, Nîmes
  - 1237.19.33019 Boehringer Ingelheim Investigational Site, Nîmes
  - 1237.19.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1237.19.33002 Boehringer Ingelheim Investigational Site, Pessac
  - 1237.19.33006 Boehringer Ingelheim Investigational Site, Reims
  - 1237.19.33021 Boehringer Ingelheim Investigational Site, Rennes
  - 1237.19.33012 Boehringer Ingelheim Investigational Site, Saint Pierre - La Réunion
  - 1237.19.33005 Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
  - 1237.19.33022 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1237.19.33007 Boehringer Ingelheim Investigational Site, Toulouse
  - 1237.19.33023 Boehringer Ingelheim Investigational Site, Tours
  - 1237.19.33010 Boehringer Ingelheim Investigational Site, Vieux-Condé
- Germany (64):
  - 1237.19.49041 Boehringer Ingelheim Investigational Site, Ahlen
  - 1237.19.49004 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1237.19.49059 Boehringer Ingelheim Investigational Site, Augsburg
  - 1237.19.49042 Boehringer Ingelheim Investigational Site, Bad Wörishofen
  - 1237.19.49072 Boehringer Ingelheim Investigational Site, Bamberg
  - 1237.19.49024 Boehringer Ingelheim Investigational Site, Bergisch Gladbach
  - 1237.19.49009 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49011 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49018 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49025 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49026 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49029 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49035 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49043 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49058 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49065 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.19.49076 Boehringer Ingelheim Investigational Site, Bielefeld
  - 1237.19.49064 Boehringer Ingelheim Investigational Site, Bochum
  - 1237.19.49048 Boehringer Ingelheim Investigational Site, Bonn
  - 1237.19.49034 Boehringer Ingelheim Investigational Site, Cologne
  - 1237.19.49002 Boehringer Ingelheim Investigational Site, Düren
  - 1237.19.49012 Boehringer Ingelheim Investigational Site, Essen
  - 1237.19.49017 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.19.49019 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.19.49052 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.19.49062 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.19.49044 Boehringer Ingelheim Investigational Site, Fulda
  - 1237.19.49057 Boehringer Ingelheim Investigational Site, Fürstenwalde
  - 1237.19.49001 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.19.49008 Boehringer Ingelheim Investigational Site, Gütersloh
  - 1237.19.49028 Boehringer Ingelheim Investigational Site, Halle
  - 1237.19.49038 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.19.49055 Boehringer Ingelheim Investigational Site, Hanover
  - 1237.19.49077 Boehringer Ingelheim Investigational Site, Hanover
  - 1237.19.49022 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1237.19.49056 Boehringer Ingelheim Investigational Site, Höchstädt
  - 1237.19.49049 Boehringer Ingelheim Investigational Site, Kiel
  - 1237.19.49005 Boehringer Ingelheim Investigational Site, Koblenz
  - 1237.19.49073 Boehringer Ingelheim Investigational Site, Landsberg am Lech
  - 1237.19.49003 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.19.49007 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.19.49030 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.19.49061 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.19.49063 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.19.49070 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.19.49010 Boehringer Ingelheim Investigational Site, Leverkusen
  - 1237.19.49037 Boehringer Ingelheim Investigational Site, Lübeck
  - 1237.19.49016 Boehringer Ingelheim Investigational Site, Mannheim
  - 1237.19.49046 Boehringer Ingelheim Investigational Site, Mannheim
  - 1237.19.49036 Boehringer Ingelheim Investigational Site, Marburg
  - 1237.19.49054 Boehringer Ingelheim Investigational Site, Minden
  - 1237.19.49006 Boehringer Ingelheim Investigational Site, München
  - 1237.19.49013 Boehringer Ingelheim Investigational Site, München
  - 1237.19.49047 Boehringer Ingelheim Investigational Site, Paderborn
  - 1237.19.49014 Boehringer Ingelheim Investigational Site, Peine
  - 1237.19.49074 Boehringer Ingelheim Investigational Site, Potsdam
  - 1237.19.49045 Boehringer Ingelheim Investigational Site, Radebeul
  - 1237.19.49053 Boehringer Ingelheim Investigational Site, Rheine
  - 1237.19.49060 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1237.19.49050 Boehringer Ingelheim Investigational Site, Solingen
  - 1237.19.49032 Boehringer Ingelheim Investigational Site, Teuchern
  - 1237.19.49051 Boehringer Ingelheim Investigational Site, Wardenburg
  - 1237.19.49040 Boehringer Ingelheim Investigational Site, Wiesloch
  - 1237.19.49023 Boehringer Ingelheim Investigational Site, Witten
- Greece (8):
  - 1237.19.30003 Boehringer Ingelheim Investigational Site, Athens
  - 1237.19.30007 Boehringer Ingelheim Investigational Site, Athens
  - 1237.19.30008 Boehringer Ingelheim Investigational Site, Athens
  - 1237.19.30004 Boehringer Ingelheim Investigational Site, Heraklion
  - 1237.19.30002 Boehringer Ingelheim Investigational Site, Nafplion
  - 1237.19.30005 Boehringer Ingelheim Investigational Site, Serres
  - 1237.19.30001 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1237.19.30006 Boehringer Ingelheim Investigational Site, Thessaloniki
- Guatemala (5):
  - 1237.19.50201 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.19.50202 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.19.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.19.50204 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1237.19.50205 Boehringer Ingelheim Investigational Site, Guatemala City
- Hong Kong (3):
  - 1237.19.85201 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1237.19.85202 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1237.19.85203 Boehringer Ingelheim Investigational Site, Hong Kong
- Hungary (15):
  - 1237.19.36006 Boehringer Ingelheim Investigational Site, Budapest
  - 1237.19.36012 Boehringer Ingelheim Investigational Site, Budapest
  - 1237.19.36005 Boehringer Ingelheim Investigational Site, Debrecen
  - 1237.19.36015 Boehringer Ingelheim Investigational Site, Debrecen
  - 1237.19.36008 Boehringer Ingelheim Investigational Site, Edelény
  - 1237.19.36011 Boehringer Ingelheim Investigational Site, Farkasgyepű
  - 1237.19.36002 Boehringer Ingelheim Investigational Site, Gödöllő
  - 1237.19.36014 Boehringer Ingelheim Investigational Site, Hajdúnánás
  - 1237.19.36013 Boehringer Ingelheim Investigational Site, Kapuvár
  - 1237.19.36009 Boehringer Ingelheim Investigational Site, Komárom
  - 1237.19.36007 Boehringer Ingelheim Investigational Site, Nyíregyháza
  - 1237.19.36003 Boehringer Ingelheim Investigational Site, Pécs
  - 1237.19.36004 Boehringer Ingelheim Investigational Site, Pécs
  - 1237.19.36010 Boehringer Ingelheim Investigational Site, Százhalombatta
  - 1237.19.36001 Boehringer Ingelheim Investigational Site, Szeged
- India (28):
  - 1237.19.91016 Boehringer Ingelheim Investigational Site, Ahmadābād
  - 1237.19.91013 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1237.19.91040 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1237.19.91032 Boehringer Ingelheim Investigational Site, Bangalore
  - 1237.19.91004 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1237.19.91033 Boehringer Ingelheim Investigational Site, Gūrgaon
  - 1237.19.91005 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1237.19.91019 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1237.19.91020 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1237.19.91025 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1237.19.91006 Boehringer Ingelheim Investigational Site, Jaipur
  - 1237.19.91042 Boehringer Ingelheim Investigational Site, Jaipur
  - 1237.19.91044 Boehringer Ingelheim Investigational Site, Jaipur
  - 1237.19.91026 Boehringer Ingelheim Investigational Site, Karamsad
  - 1237.19.91034 Boehringer Ingelheim Investigational Site, Kolkata
  - 1237.19.91010 Boehringer Ingelheim Investigational Site, Ludhiana
  - 1237.19.91007 Boehringer Ingelheim Investigational Site, Madurai
  - 1237.19.91014 Boehringer Ingelheim Investigational Site, Mysore
  - 1237.19.91021 Boehringer Ingelheim Investigational Site, Mysore
  - 1237.19.91001 Boehringer Ingelheim Investigational Site, Nagpur
  - 1237.19.91002 Boehringer Ingelheim Investigational Site, Nagpur
  - 1237.19.91003 Boehringer Ingelheim Investigational Site, Nagpur
  - 1237.19.91027 Boehringer Ingelheim Investigational Site, New Delhi
  - 1237.19.91024 Boehringer Ingelheim Investigational Site, Panjim
  - 1237.19.91023 Boehringer Ingelheim Investigational Site, Pune
  - 1237.19.91035 Boehringer Ingelheim Investigational Site, Pune
  - 1237.19.91008 Boehringer Ingelheim Investigational Site, Vellore
  - 1237.19.91028 Boehringer Ingelheim Investigational Site, Visakhapatnam
- Ireland (2):
  - 1237.19.35301 Boehringer Ingelheim Investigational Site, Dublin
  - 1237.19.35302 Boehringer Ingelheim Investigational Site, Wilton
- Italy (22):
  - 1237.19.39011 Boehringer Ingelheim Investigational Site, Cittadella (PD)
  - 1237.19.39014 Boehringer Ingelheim Investigational Site, Ferrara
  - 1237.19.39010 Boehringer Ingelheim Investigational Site, Messina
  - 1237.19.39002 Boehringer Ingelheim Investigational Site, Milan
  - 1237.19.39016 Boehringer Ingelheim Investigational Site, Milan
  - 1237.19.39023 Boehringer Ingelheim Investigational Site, Milan
  - 1237.19.39015 Boehringer Ingelheim Investigational Site, Monza
  - 1237.19.39025 Boehringer Ingelheim Investigational Site, Padua
  - 1237.19.39024 Boehringer Ingelheim Investigational Site, Palermo
  - 1237.19.39006 Boehringer Ingelheim Investigational Site, Parma
  - 1237.19.39005 Boehringer Ingelheim Investigational Site, Pavia
  - 1237.19.39007 Boehringer Ingelheim Investigational Site, Perugia
  - 1237.19.39008 Boehringer Ingelheim Investigational Site, Piacenza
  - 1237.19.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1237.19.39020 Boehringer Ingelheim Investigational Site, Pisa
  - 1237.19.39013 Boehringer Ingelheim Investigational Site, Pordenone
  - 1237.19.39003 Boehringer Ingelheim Investigational Site, Roma
  - 1237.19.39004 Boehringer Ingelheim Investigational Site, Roma
  - 1237.19.39012 Boehringer Ingelheim Investigational Site, Roma
  - 1237.19.39021 Boehringer Ingelheim Investigational Site, San Pietro Vernotico (BR)
  - 1237.19.39017 Boehringer Ingelheim Investigational Site, Sassari
  - 1237.19.39019 Boehringer Ingelheim Investigational Site, Scafati (SA)
- Japan (124):
  - 1237.19.81072 Boehringer Ingelheim Investigational Site, Aichi, Komaki
  - 1237.19.81070 Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - 1237.19.81073 Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - 1237.19.81074 Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - 1237.19.81071 Boehringer Ingelheim Investigational Site, Aichi, Obu
  - 1237.19.81069 Boehringer Ingelheim Investigational Site, Aichi, Seto
  - 1237.19.81030 Boehringer Ingelheim Investigational Site, Chiba, Chiba
  - 1237.19.81031 Boehringer Ingelheim Investigational Site, Chiba, Kamogawa
  - 1237.19.81061 Boehringer Ingelheim Investigational Site, Fukui, Fukui
  - 1237.19.81116 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1237.19.81112 Boehringer Ingelheim Investigational Site, Fukuoka, Kitakyushu-city
  - 1237.19.81113 Boehringer Ingelheim Investigational Site, Fukuoka, Koga
  - 1237.19.81111 Boehringer Ingelheim Investigational Site, Fukuoka, Kurume
  - 1237.19.81114 Boehringer Ingelheim Investigational Site, Fukuoka, Yanagawa
  - 1237.19.81115 Boehringer Ingelheim Investigational Site, Fukuoka, Yukuhashi
  - 1237.19.81022 Boehringer Ingelheim Investigational Site, Fukushima, Fukushima
  - 1237.19.81066 Boehringer Ingelheim Investigational Site, Gifu, Mizunami
  - 1237.19.81065 Boehringer Ingelheim Investigational Site, Gifu, Ogaki
  - 1237.19.81025 Boehringer Ingelheim Investigational Site, Gunma, Fujioka
  - 1237.19.81027 Boehringer Ingelheim Investigational Site, Gunma, Maebashi
  - 1237.19.81026 Boehringer Ingelheim Investigational Site, Gunma, Takasaki
  - 1237.19.81101 Boehringer Ingelheim Investigational Site, Hiroshima, Fukuyama
  - 1237.19.81104 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 1237.19.81102 Boehringer Ingelheim Investigational Site, Hiroshima, Kure
  - 1237.19.81103 Boehringer Ingelheim Investigational Site, Hiroshima, Kure
  - 1237.19.81010 Boehringer Ingelheim Investigational Site, Hokkaido, Asahikawa
  - 1237.19.81007 Boehringer Ingelheim Investigational Site, Hokkaido, Chitose
  - 1237.19.81012 Boehringer Ingelheim Investigational Site, Hokkaido, Hakodate
  - 1237.19.81013 Boehringer Ingelheim Investigational Site, Hokkaido, Hakodate
  - 1237.19.81009 Boehringer Ingelheim Investigational Site, Hokkaido, Obihiro
  - 1237.19.81015 Boehringer Ingelheim Investigational Site, Hokkaido, Obihiro
  - 1237.19.81016 Boehringer Ingelheim Investigational Site, Hokkaido, Otaru
  - 1237.19.81001 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81002 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81004 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81006 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81008 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81011 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81014 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81017 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1237.19.81003 Boehringer Ingelheim Investigational Site, Hokkaido, Tomakomai
  - 1237.19.81090 Boehringer Ingelheim Investigational Site, Hyogo, Himeji
  - 1237.19.81093 Boehringer Ingelheim Investigational Site, Hyogo, Himeji
  - 1237.19.81091 Boehringer Ingelheim Investigational Site, Hyogo, Kobe
  - 1237.19.81092 Boehringer Ingelheim Investigational Site, Hyogo, Nishinomiya
  - 1237.19.81024 Boehringer Ingelheim Investigational Site, Ibaraki, Hitachinaka
  - 1237.19.81129 Boehringer Ingelheim Investigational Site, Ibaraki, Inashiki-gun
  - 1237.19.81023 Boehringer Ingelheim Investigational Site, Ibaraki, Naka-gun
  - 1237.19.81060 Boehringer Ingelheim Investigational Site, Ishikawa, Kanazawa
  - 1237.19.81018 Boehringer Ingelheim Investigational Site, Iwate, Morioka
  - 1237.19.81108 Boehringer Ingelheim Investigational Site, Kagawa, Sakaide
  - 1237.19.81107 Boehringer Ingelheim Investigational Site, Kagawa, Takamatsu
  - 1237.19.81109 Boehringer Ingelheim Investigational Site, Kagawa, Takamatsu
  - 1237.19.81118 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima
  - 1237.19.81050 Boehringer Ingelheim Investigational Site, Kanagawa, Isehara
  - 1237.19.81052 Boehringer Ingelheim Investigational Site, Kanagawa, Kawasaki
  - 1237.19.81053 Boehringer Ingelheim Investigational Site, Kanagawa, Kawasaki
  - 1237.19.81055 Boehringer Ingelheim Investigational Site, Kanagawa, Kawasaki
  - 1237.19.81054 Boehringer Ingelheim Investigational Site, Kanagawa, Sagamihara
  - 1237.19.81056 Boehringer Ingelheim Investigational Site, Kanagawa, Sagamihara
  - 1237.19.81049 Boehringer Ingelheim Investigational Site, Kanagawa, Yokohama
  - 1237.19.81051 Boehringer Ingelheim Investigational Site, Kanagawa, Yokohama
  - 1237.19.81110 Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - 1237.19.81130 Boehringer Ingelheim Investigational Site, Kochi, Nankoku
  - 1237.19.81077 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1237.19.81076 Boehringer Ingelheim Investigational Site, Mie, Matsusaka
  - 1237.19.81005 Boehringer Ingelheim Investigational Site, Miyagi, Sendai
  - 1237.19.81019 Boehringer Ingelheim Investigational Site, Miyagi, Sendai
  - 1237.19.81020 Boehringer Ingelheim Investigational Site, Miyagi, Sendai
  - 1237.19.81038 Boehringer Ingelheim Investigational Site, Miyagi, Sendai
  - 1237.19.81064 Boehringer Ingelheim Investigational Site, Nagano, Matsumoto
  - 1237.19.81063 Boehringer Ingelheim Investigational Site, Nagano, Matumoto
  - 1237.19.81117 Boehringer Ingelheim Investigational Site, Nagasaki, Isahaya
  - 1237.19.81095 Boehringer Ingelheim Investigational Site, Nara, Ikoma
  - 1237.19.81057 Boehringer Ingelheim Investigational Site, Niigata, Niigata
  - 1237.19.81058 Boehringer Ingelheim Investigational Site, Niigata, Niigata
  - 1237.19.81059 Boehringer Ingelheim Investigational Site, Niigata, Niigata
  - 1237.19.81125 Boehringer Ingelheim Investigational Site, Okayama
  - 1237.19.81100 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1237.19.81119 Boehringer Ingelheim Investigational Site, Okinawa, Urasoe
  - 1237.19.81120 Boehringer Ingelheim Investigational Site, Okinawa, Uruma
  - 1237.19.81089 Boehringer Ingelheim Investigational Site, Osaka, Ikeda
  - 1237.19.81082 Boehringer Ingelheim Investigational Site, Osaka, Kishiwada
  - 1237.19.81078 Boehringer Ingelheim Investigational Site, Osaka, Osakasayama
  - 1237.19.81079 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1237.19.81080 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1237.19.81086 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1237.19.81088 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1237.19.81083 Boehringer Ingelheim Investigational Site, Osaka, Sakai
  - 1237.19.81081 Boehringer Ingelheim Investigational Site, Osaka, Takatsuki
  - 1237.19.81085 Boehringer Ingelheim Investigational Site, Osaka, Toyonaka
  - 1237.19.81087 Boehringer Ingelheim Investigational Site, Osaka, Yao
  - 1237.19.81028 Boehringer Ingelheim Investigational Site, Saitama, Koshigaya
  - 1237.19.81029 Boehringer Ingelheim Investigational Site, Saitama, Saitama
  - 1237.19.81128 Boehringer Ingelheim Investigational Site, Shiga
  - 1237.19.81098 Boehringer Ingelheim Investigational Site, Shimane, Izumo
  - 1237.19.81099 Boehringer Ingelheim Investigational Site, Shimane, Izumo
  - 1237.19.81067 Boehringer Ingelheim Investigational Site, Shizuoka, Hamamatsu
  - 1237.19.81068 Boehringer Ingelheim Investigational Site, Shizuoka, Shizuoka
  - 1237.19.81123 Boehringer Ingelheim Investigational Site, Tochigi, Shimotsuke
  - 1237.19.81122 Boehringer Ingelheim Investigational Site, Tokyo
  - 1237.19.81126 Boehringer Ingelheim Investigational Site, Tokyo
  - 1237.19.81075 Boehringer Ingelheim Investigational Site, Tokyo, Chiyoda-ku
  - 1237.19.81036 Boehringer Ingelheim Investigational Site, Tokyo, Chuo-ku
  - 1237.19.81040 Boehringer Ingelheim Investigational Site, Tokyo, Chuo-ku
  - 1237.19.81039 Boehringer Ingelheim Investigational Site, Tokyo, Hachioji
  - 1237.19.81035 Boehringer Ingelheim Investigational Site, Tokyo, Itabashi-ku
  - 1237.19.81043 Boehringer Ingelheim Investigational Site, Tokyo, Itabashi-ku
  - 1237.19.81046 Boehringer Ingelheim Investigational Site, Tokyo, Koto-ku
  - 1237.19.81034 Boehringer Ingelheim Investigational Site, Tokyo, Meguro-ku
  - 1237.19.81032 Boehringer Ingelheim Investigational Site, Tokyo, Minato-ku
  - 1237.19.81047 Boehringer Ingelheim Investigational Site, Tokyo, Shinagawa-ku
  - 1237.19.81033 Boehringer Ingelheim Investigational Site, Tokyo, Shinjuku-ku
  - 1237.19.81041 Boehringer Ingelheim Investigational Site, Tokyo, Shinjuku-ku
  - 1237.19.81042 Boehringer Ingelheim Investigational Site, Tokyo, Shinjuku-ku
  - 1237.19.81044 Boehringer Ingelheim Investigational Site, Tokyo, Tachikawa
  - 1237.19.81048 Boehringer Ingelheim Investigational Site, Tokyo, Toshima-ku
  - 1237.19.81097 Boehringer Ingelheim Investigational Site, Wakayama, Hidaka-gun
  - 1237.19.81096 Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
  - 1237.19.81124 Boehringer Ingelheim Investigational Site, Yamagata
  - 1237.19.81021 Boehringer Ingelheim Investigational Site, Yamagata, Yonezawa
  - 1237.19.81106 Boehringer Ingelheim Investigational Site, Yamaguchi, Iwakuni
  - 1237.19.81105 Boehringer Ingelheim Investigational Site, Yamaguchi, Ube
  - 1237.19.81062 Boehringer Ingelheim Investigational Site, Yamanashi, Kofu
- Latvia (6):
  - 1237.19.37103 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1237.19.37101 Boehringer Ingelheim Investigational Site, Riga
  - 1237.19.37105 Boehringer Ingelheim Investigational Site, Riga
  - 1237.19.37106 Boehringer Ingelheim Investigational Site, Riga
  - 1237.19.37104 Boehringer Ingelheim Investigational Site, Tukums
  - 1237.19.37102 Boehringer Ingelheim Investigational Site, Valmiera
- Lithuania (4):
  - 1237.19.37002 Boehringer Ingelheim Investigational Site, Kaunas
  - 1237.19.37003 Boehringer Ingelheim Investigational Site, Klaipėda
  - 1237.19.37004 Boehringer Ingelheim Investigational Site, Klaipėda
  - 1237.19.37001 Boehringer Ingelheim Investigational Site, Vilnius
- Malaysia (4):
  - 1237.19.60006 Boehringer Ingelheim Investigational Site, Kota Bharu
  - 1237.19.60002 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1237.19.60004 Boehringer Ingelheim Investigational Site, Kuala Terengganu
  - 1237.19.60001 Boehringer Ingelheim Investigational Site, Kuching
- Mexico (6):
  - 1237.19.52006 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1237.19.52007 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1237.19.52005 Boehringer Ingelheim Investigational Site, León
  - 1237.19.52003 Boehringer Ingelheim Investigational Site, México
  - 1237.19.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1237.19.52004 Boehringer Ingelheim Investigational Site, Tijuana
- Netherlands (16):
  - 1237.19.31017 Boehringer Ingelheim Investigational Site, Alkmaar
  - 1237.19.31015 Boehringer Ingelheim Investigational Site, Almelo
  - 1237.19.31011 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1237.19.31014 Boehringer Ingelheim Investigational Site, Assen
  - 1237.19.31001 Boehringer Ingelheim Investigational Site, Breda
  - 1237.19.31003 Boehringer Ingelheim Investigational Site, Ede
  - 1237.19.31002 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1237.19.31005 Boehringer Ingelheim Investigational Site, Groningen
  - 1237.19.31010 Boehringer Ingelheim Investigational Site, Harderwijk
  - 1237.19.31012 Boehringer Ingelheim Investigational Site, Hoofddorp
  - 1237.19.31013 Boehringer Ingelheim Investigational Site, Hoorn
  - 1237.19.31018 Boehringer Ingelheim Investigational Site, Leeuwarden
  - 1237.19.31016 Boehringer Ingelheim Investigational Site, Leiden
  - 1237.19.31008 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1237.19.31007 Boehringer Ingelheim Investigational Site, Sittard - Geleen
  - 1237.19.31004 Boehringer Ingelheim Investigational Site, Zutphen
- New Zealand (8):
  - 1237.19.64003 Boehringer Ingelheim Investigational Site, Auckland, New Zealand
  - 1237.19.64002 Boehringer Ingelheim Investigational Site, Christchurch
  - 1237.19.64004 Boehringer Ingelheim Investigational Site, Christchurch Central
  - 1237.19.64007 Boehringer Ingelheim Investigational Site, Dunedin
  - 1237.19.64008 Boehringer Ingelheim Investigational Site, Dunedin
  - 1237.19.64001 Boehringer Ingelheim Investigational Site, Greenlane East Auckland NZ
  - 1237.19.64005 Boehringer Ingelheim Investigational Site, Hamilton
  - 1237.19.64009 Boehringer Ingelheim Investigational Site, Tauranga
- Norway (7):
  - 1237.19.47002 Boehringer Ingelheim Investigational Site, Arendal
  - 1237.19.47008 Boehringer Ingelheim Investigational Site, Hamar
  - 1237.19.47001 Boehringer Ingelheim Investigational Site, Hønefoss
  - 1237.19.47006 Boehringer Ingelheim Investigational Site, Kløfta
  - 1237.19.47007 Boehringer Ingelheim Investigational Site, Lierskogen
  - 1237.19.47004 Boehringer Ingelheim Investigational Site, Oslo
  - 1237.19.47005 Boehringer Ingelheim Investigational Site, Skedsmokorset
- Philippines (7):
  - 1237.19.63007 Boehringer Ingelheim Investigational Site, Angeles City
  - 1237.19.63001 Boehringer Ingelheim Investigational Site, Cebu City
  - 1237.19.63003 Boehringer Ingelheim Investigational Site, Dasmariñas
  - 1237.19.63008 Boehringer Ingelheim Investigational Site, Davao City
  - 1237.19.63006 Boehringer Ingelheim Investigational Site, Iloilo City
  - 1237.19.63005 Boehringer Ingelheim Investigational Site, Manila
  - 1237.19.63002 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (29):
  - 1237.19.48009 Boehringer Ingelheim Investigational Site, Bialystok
  - 1237.19.48026 Boehringer Ingelheim Investigational Site, Bialystok
  - 1237.19.48031 Boehringer Ingelheim Investigational Site, Bialystok
  - 1237.19.48010 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1237.19.48029 Boehringer Ingelheim Investigational Site, Chojnice
  - 1237.19.48001 Boehringer Ingelheim Investigational Site, Katowice
  - 1237.19.48024 Boehringer Ingelheim Investigational Site, Kielce
  - 1237.19.48005 Boehringer Ingelheim Investigational Site, Krakow
  - 1237.19.48007 Boehringer Ingelheim Investigational Site, Krakow
  - 1237.19.48015 Boehringer Ingelheim Investigational Site, Libiąż
  - 1237.19.48006 Boehringer Ingelheim Investigational Site, Lodz
  - 1237.19.48008 Boehringer Ingelheim Investigational Site, Lodz
  - 1237.19.48025 Boehringer Ingelheim Investigational Site, Lublin
  - 1237.19.48011 Boehringer Ingelheim Investigational Site, Olsztyn
  - 1237.19.48013 Boehringer Ingelheim Investigational Site, Ostow Wielkopolski
  - 1237.19.48019 Boehringer Ingelheim Investigational Site, Ostróda
  - 1237.19.48020 Boehringer Ingelheim Investigational Site, Piaseczno
  - 1237.19.48002 Boehringer Ingelheim Investigational Site, Poznan
  - 1237.19.48004 Boehringer Ingelheim Investigational Site, Poznan
  - 1237.19.48014 Boehringer Ingelheim Investigational Site, Poznan
  - 1237.19.48016 Boehringer Ingelheim Investigational Site, Skierniewice
  - 1237.19.48017 Boehringer Ingelheim Investigational Site, Szczecin
  - 1237.19.48021 Boehringer Ingelheim Investigational Site, Świdnik
  - 1237.19.48030 Boehringer Ingelheim Investigational Site, Tarnobrzeg
  - 1237.19.48022 Boehringer Ingelheim Investigational Site, Warsaw
  - 1237.19.48003 Boehringer Ingelheim Investigational Site, Wołomin
  - 1237.19.48023 Boehringer Ingelheim Investigational Site, Wroclaw
  - 1237.19.48018 Boehringer Ingelheim Investigational Site, Zawadzkie
  - 1237.19.48012 Boehringer Ingelheim Investigational Site, Zgierz
- Portugal (10):
  - 1237.19.35010 Boehringer Ingelheim Investigational Site, Almada
  - 1237.19.35005 Boehringer Ingelheim Investigational Site, Amadora
  - 1237.19.35008 Boehringer Ingelheim Investigational Site, Aveiro
  - 1237.19.35009 Boehringer Ingelheim Investigational Site, Braga
  - 1237.19.35001 Boehringer Ingelheim Investigational Site, Coimbra
  - 1237.19.35012 Boehringer Ingelheim Investigational Site, Guimarães
  - 1237.19.35002 Boehringer Ingelheim Investigational Site, Lisbon
  - 1237.19.35004 Boehringer Ingelheim Investigational Site, Lisbon
  - 1237.19.35003 Boehringer Ingelheim Investigational Site, Porto
  - 1237.19.35006 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
- Romania (7):
  - 1237.19.40007 Boehringer Ingelheim Investigational Site, Bragadiru
  - 1237.19.40003 Boehringer Ingelheim Investigational Site, Bucharest
  - 1237.19.40004 Boehringer Ingelheim Investigational Site, Bucharest
  - 1237.19.40005 Boehringer Ingelheim Investigational Site, Bucharest
  - 1237.19.40008 Boehringer Ingelheim Investigational Site, Bucharest
  - 1237.19.40002 Boehringer Ingelheim Investigational Site, Constanța
  - 1237.19.40006 Boehringer Ingelheim Investigational Site, Timișoara
- Russia (44):
  - 1237.19.70004 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 1237.19.70028 Boehringer Ingelheim Investigational Site, Barnaul
  - 1237.19.70017 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1237.19.70014 Boehringer Ingelheim Investigational Site, Gatchina
  - 1237.19.70051 Boehringer Ingelheim Investigational Site, Ivanovo
  - 1237.19.70050 Boehringer Ingelheim Investigational Site, Kazan'
  - 1237.19.70006 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1237.19.70023 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1237.19.70031 Boehringer Ingelheim Investigational Site, Kirov
  - 1237.19.70007 Boehringer Ingelheim Investigational Site, Lomonosov
  - 1237.19.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.19.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.19.70032 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.19.70047 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.19.70024 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1237.19.70025 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1237.19.70034 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1237.19.70035 Boehringer Ingelheim Investigational Site, Omsk
  - 1237.19.70033 Boehringer Ingelheim Investigational Site, Penza
  - 1237.19.70021 Boehringer Ingelheim Investigational Site, Pskov
  - 1237.19.70052 Boehringer Ingelheim Investigational Site, Rosto-on-Don
  - 1237.19.70015 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1237.19.70009 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70010 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70011 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70012 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70018 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70019 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70022 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70038 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70041 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70042 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70046 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70048 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70049 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.19.70005 Boehringer Ingelheim Investigational Site, Saratov
  - 1237.19.70040 Boehringer Ingelheim Investigational Site, Saratov
  - 1237.19.70044 Boehringer Ingelheim Investigational Site, Saratov
  - 1237.19.70008 Boehringer Ingelheim Investigational Site, Tomsk
  - 1237.19.70026 Boehringer Ingelheim Investigational Site, Tomsk
  - 1237.19.70037 Boehringer Ingelheim Investigational Site, Ulyanovsk
  - 1237.19.70030 Boehringer Ingelheim Investigational Site, Volgograd
  - 1237.19.70036 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1237.19.70020 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Serbia (8):
  - 1237.19.38101 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.19.38102 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.19.38105 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.19.38107 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.19.38103 Boehringer Ingelheim Investigational Site, Kamenitz
  - 1237.19.38104 Boehringer Ingelheim Investigational Site, Kragujevac
  - 1237.19.38108 Boehringer Ingelheim Investigational Site, Niš
  - 1237.19.38106 Boehringer Ingelheim Investigational Site, Sombor
- Singapore (2):
  - 1237.19.65001 Boehringer Ingelheim Investigational Site, Singapore
  - 1237.19.65002 Boehringer Ingelheim Investigational Site, Singapore
- Slovakia (7):
  - 1237.19.42101 Boehringer Ingelheim Investigational Site, Bratislava
  - 1237.19.42104 Boehringer Ingelheim Investigational Site, Humenné
  - 1237.19.42102 Boehringer Ingelheim Investigational Site, Košice
  - 1237.19.42106 Boehringer Ingelheim Investigational Site, Martin
  - 1237.19.42107 Boehringer Ingelheim Investigational Site, Poprad
  - 1237.19.42103 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
  - 1237.19.42105 Boehringer Ingelheim Investigational Site, Vráble
- Slovenia (3):
  - 1237.19.38601 Boehringer Ingelheim Investigational Site, Golnik
  - 1237.19.38603 Boehringer Ingelheim Investigational Site, Pohorje
  - 1237.19.38602 Boehringer Ingelheim Investigational Site, Topolšica
- South Africa (10):
  - 1237.19.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.19.27002 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.19.27003 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.19.27007 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.19.27009 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.19.27006 Boehringer Ingelheim Investigational Site, eManzimtoti
  - 1237.19.27011 Boehringer Ingelheim Investigational Site, Morningside, Sandton
  - 1237.19.27010 Boehringer Ingelheim Investigational Site, Parow
  - 1237.19.27004 Boehringer Ingelheim Investigational Site, Pretoria
  - 1237.19.27008 Boehringer Ingelheim Investigational Site, Pretoria
- South Korea (10):
  - 1237.19.82004 Boehringer Ingelheim Investigational Site, Bucheon-si
  - 1237.19.82009 Boehringer Ingelheim Investigational Site, Goyang
  - 1237.19.82006 Boehringer Ingelheim Investigational Site, Gwangju
  - 1237.19.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.19.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.19.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.19.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.19.82008 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.19.82010 Boehringer Ingelheim Investigational Site, Seoul
  - 1237.19.82003 Boehringer Ingelheim Investigational Site, Wŏnju
- Spain (26):
  - 1237.19.34017 Boehringer Ingelheim Investigational Site, Alicante
  - 1237.19.34025 Boehringer Ingelheim Investigational Site, Aranjuez
  - 1237.19.34024 Boehringer Ingelheim Investigational Site, Badalona
  - 1237.19.34011 Boehringer Ingelheim Investigational Site, Barakaldo (Bilbao)
  - 1237.19.34012 Boehringer Ingelheim Investigational Site, Barcelona
  - 1237.19.34021 Boehringer Ingelheim Investigational Site, Barcelona
  - 1237.19.34007 Boehringer Ingelheim Investigational Site, Cáceres
  - 1237.19.34028 Boehringer Ingelheim Investigational Site, Centelles
  - 1237.19.34015 Boehringer Ingelheim Investigational Site, Girona
  - 1237.19.34027 Boehringer Ingelheim Investigational Site, Granollers (Barcelona)
  - 1237.19.34003 Boehringer Ingelheim Investigational Site, L'Hospitalet Llobregat (bcn)
  - 1237.19.34001 Boehringer Ingelheim Investigational Site, Liencres (Pielagos)
  - 1237.19.34005 Boehringer Ingelheim Investigational Site, Madrid
  - 1237.19.34020 Boehringer Ingelheim Investigational Site, Madrid
  - 1237.19.34009 Boehringer Ingelheim Investigational Site, Málaga
  - 1237.19.34019 Boehringer Ingelheim Investigational Site, Mérida
  - 1237.19.34013 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1237.19.34004 Boehringer Ingelheim Investigational Site, Pamplona
  - 1237.19.34018 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 1237.19.34023 Boehringer Ingelheim Investigational Site, Sabadell
  - 1237.19.34014 Boehringer Ingelheim Investigational Site, Seville
  - 1237.19.34006 Boehringer Ingelheim Investigational Site, Valencia
  - 1237.19.34029 Boehringer Ingelheim Investigational Site, Valladolid
  - 1237.19.34026 Boehringer Ingelheim Investigational Site, Vic
  - 1237.19.34022 Boehringer Ingelheim Investigational Site, Vilanova i la Geltrú
  - 1237.19.34002 Boehringer Ingelheim Investigational Site, Zaragoza
- Sweden (6):
  - 1237.19.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1237.19.46008 Boehringer Ingelheim Investigational Site, Härnösand
  - 1237.19.46004 Boehringer Ingelheim Investigational Site, Höllviken
  - 1237.19.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1237.19.46005 Boehringer Ingelheim Investigational Site, Rättvik
  - 1237.19.46007 Boehringer Ingelheim Investigational Site, Stockholm
- Switzerland (3):
  - 1237.19.41004 Boehringer Ingelheim Investigational Site, Ascona
  - 1237.19.41002 Boehringer Ingelheim Investigational Site, Bern
  - 1237.19.41001 Boehringer Ingelheim Investigational Site, Liestal
- Taiwan (10):
  - 1237.19.88010 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1237.19.88011 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1237.19.88012 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1237.19.88004 Boehringer Ingelheim Investigational Site, New Taipei City
  - 1237.19.88009 Boehringer Ingelheim Investigational Site, New Taipei City
  - 1237.19.88001 Boehringer Ingelheim Investigational Site, Taipei
  - 1237.19.88005 Boehringer Ingelheim Investigational Site, Taipei
  - 1237.19.88007 Boehringer Ingelheim Investigational Site, Taipei
  - 1237.19.88008 Boehringer Ingelheim Investigational Site, Taipei
  - 1237.19.88013 Boehringer Ingelheim Investigational Site, Taipei
- Thailand (7):
  - 1237.19.66008 Boehringer Ingelheim Investigational Site, Dusit
  - 1237.19.66005 Boehringer Ingelheim Investigational Site, Hat Yai
  - 1237.19.66003 Boehringer Ingelheim Investigational Site, Maerim
  - 1237.19.66001 Boehringer Ingelheim Investigational Site, Muang
  - 1237.19.66002 Boehringer Ingelheim Investigational Site, Muang
  - 1237.19.66007 Boehringer Ingelheim Investigational Site, Patumwan
  - 1237.19.66004 Boehringer Ingelheim Investigational Site, Rajathevee
- Turkey (Türkiye) (17):
  - 1237.19.90006 Boehringer Ingelheim Investigational Site, Ankara
  - 1237.19.90007 Boehringer Ingelheim Investigational Site, Ankara
  - 1237.19.90015 Boehringer Ingelheim Investigational Site, Ankara
  - 1237.19.90016 Boehringer Ingelheim Investigational Site, Ankara
  - 1237.19.90008 Boehringer Ingelheim Investigational Site, Antalya
  - 1237.19.90010 Boehringer Ingelheim Investigational Site, Bursa
  - 1237.19.90002 Boehringer Ingelheim Investigational Site, Denizli
  - 1237.19.90012 Boehringer Ingelheim Investigational Site, Istanbul
  - 1237.19.90013 Boehringer Ingelheim Investigational Site, Istanbul
  - 1237.19.90014 Boehringer Ingelheim Investigational Site, Istanbul
  - 1237.19.90003 Boehringer Ingelheim Investigational Site, Izmir
  - 1237.19.90004 Boehringer Ingelheim Investigational Site, Izmir
  - 1237.19.90005 Boehringer Ingelheim Investigational Site, Izmir
  - 1237.19.90011 Boehringer Ingelheim Investigational Site, Izmir
  - 1237.19.90001 Boehringer Ingelheim Investigational Site, Kocaeli
  - 1237.19.90009 Boehringer Ingelheim Investigational Site, Konya
  - 1237.19.90000 Boehringer Ingelheim Investigational Site, Mersin
- Ukraine (10):
  - 1237.19.38009 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 1237.19.38001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1237.19.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 1237.19.38007 Boehringer Ingelheim Investigational Site, Kiev
  - 1237.19.38002 Boehringer Ingelheim Investigational Site, Kyiv
  - 1237.19.38003 Boehringer Ingelheim Investigational Site, Kyiv
  - 1237.19.38004 Boehringer Ingelheim Investigational Site, Kyiv
  - 1237.19.38006 Boehringer Ingelheim Investigational Site, Kyiv
  - 1237.19.38010 Boehringer Ingelheim Investigational Site, Odesa
  - 1237.19.38008 Boehringer Ingelheim Investigational Site, Vinnytsia
- United Kingdom (7):
  - 1237.19.44008 Boehringer Ingelheim Investigational Site, Bedford
  - 1237.19.44006 Boehringer Ingelheim Investigational Site, Birmingham
  - 1237.19.44001 Boehringer Ingelheim Investigational Site, Bradford
  - 1237.19.44002 Boehringer Ingelheim Investigational Site, Chertsey
  - 1237.19.44004 Boehringer Ingelheim Investigational Site, Coventry
  - 1237.19.44007 Boehringer Ingelheim Investigational Site, Doncaster
  - 1237.19.44003 Boehringer Ingelheim Investigational Site, South Shields
- Vietnam (3):
  - 1237.19.84003 Boehringer Ingelheim Investigational Site, Hà Nội
  - 1237.19.84001 Boehringer Ingelheim Investigational Site, Ho Chi Minh City
  - 1237.19.84002 Boehringer Ingelheim Investigational Site, Ho Chi Minh City

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Wedzicha JA, Buhl R, Singh D, Vogelmeier CF, de la Hoz A, Xue W, Anzueto A, Calverley PMA. Tiotropium/Olodaterol Decreases Exacerbation Rates Compared with Tiotropium in a Range of Patients with COPD: Pooled Analysis of the TONADO(R)/DYNAGITO(R) Trials. Adv Ther. 2020 Oct;37(10):4266-4279. doi: 10.1007/s12325-020-01438-3. Epub 2020 Aug 10. PMID 32776202
- [Derived] Ferguson GT, Buhl R, Bothner U, Hoz A, Voss F, Anzueto A, Calverley PMA. Safety of tiotropium/olodaterol in chronic obstructive pulmonary disease: pooled analysis of three large, 52-week, randomized clinical trials. Respir Med. 2018 Oct;143:67-73. doi: 10.1016/j.rmed.2018.08.012. Epub 2018 Aug 28. PMID 30261995
- [Derived] Calverley PMA, Anzueto AR, Carter K, Gronke L, Hallmann C, Jenkins C, Wedzicha J, Rabe KF. Tiotropium and olodaterol in the prevention of chronic obstructive pulmonary disease exacerbations (DYNAGITO): a double-blind, randomised, parallel-group, active-controlled trial. Lancet Respir Med. 2018 May;6(5):337-344. doi: 10.1016/S2213-2600(18)30102-4. Epub 2018 Apr 5. PMID 29605624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, double-blind, active-controlled parallel group study to evaluate the effect of 52 weeks of once daily treatment of orally inhaled tiotropium + olodaterol fixed dose combination compared with tiotropium on Chronic Obstructive Pulmonary Disease (COPD) exacerbation in patients with severe to very severe COPD.
Pre-assignment Details: Following informed consent, the patient was entered into a maximum 7-day screening period to confirm the patient's eligibility. At Visit 2, after a successful review of the inclusion and exclusion criteria, the patient was randomly allocated in equal ratio to receive once daily trial treatment and then entered the 360 days treatment phase.
Groups:
- Tiotropium 5 Microgram (μg): Patient received 5 μg Tiotropium inhalation solution - RESPIMAT inhaler once daily orally for 360 days
- Tiotropium (5 μg) + Olodaterol (5 μg): Patient received 5 μg Tiotropium + 5 μg Olodaterol fixed-dose combination (FDC) inhalation solution - RESPIMAT inhaler once daily orally for 360 days
Period: Overall Study
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
Started | 3952 | 3951
Treated | 3941 | 3939
Completed | 3291 | 3451
Not Completed | 661 | 500
Not completed — Adverse Event | 348 | 259
Not completed — Lack of Efficacy | 59 | 37
Not completed — Protocol Violation | 35 | 36
Not completed — Lost to Follow-up | 9 | 12
Not completed — Withdrawal by Subject | 184 | 131
Not completed — Not Treated | 1 | 1
Not completed — Patients with data irregularities | 10 | 11
Not completed — Other than specified | 15 | 13

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set includes all randomised patients who were documented to have taken at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg) | Total
Number analyzed (Participants) | 3941 | 3939 | 7880
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: Treated Set
  Years | 66.3 (8.5) | 66.5 (8.4) | 66.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: Treated Set
  Participants
    Female | 1100 | 1154 | 2254
    Male | 2841 | 2785 | 5626
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not captured in this trial Population: Treated Set
  Participants
    American Indian or Alaska Native | 64 | 77 | 141
    Asian | 607 | 557 | 1164
    Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
    Black or African American | 52 | 58 | 110
    White | 3113 | 3134 | 6247
    More than one race | 20 | 22 | 42
    Unknown or Not Reported | 80 | 88 | 168

OUTCOME MEASURES:

1. Primary Outcome: Annualised Rate of Moderate to Severe COPD Exacerbations During the Actual Treatment Period.
Description: Annualised rate of moderate to severe COPD exacerbations during the actual treatment period was calculated per treatment per patient-year. The actual treatment period was defined as the interval from first in-take of study medication until 1 day after last in-take of study medication. Least Squares Means are actually exponentiated.
Time Frame: From first in-take of study medication until 1 day after last in-take of study medication, up to 361 days
Population: Treated set (TS) -This patient set includes all randomised patients who were documented to have taken at least 1 dose of trial medication.
Measure: Least Squares Mean (99% Confidence Interval); unit: Rate per patient-year
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
Number analyzed (Participants) | 3941 | 3939
Rate per patient-year | 0.97 [0.90 to 1.03] | 0.90 [0.84 to 0.96]
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); Annualised rate of moderate to severe COPD exacerbation was analysed using a negative binomial model including the fixed, categorical effect of treatment as well as the logarithm of the treatment exposure as an offset; Test type: Superiority — This hypothesis testing strategy ensures that the overall type I error is protected at 2-sided 0.01 level; p = 0.0498, Negative binomial model; Ratio of rates vs. Tiotropium 5 μg = 0.93, 99% CI 2-sided [0.85 to 1.02] — Ratio of events Tiotropium (5 μg) + Olodaterol (5 μg) versus Tiotropium (5 μg) is provided
Statistical Analysis 2: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); Model was based on SPARK/FLAME- Covariates: Smoking status, baseline inhaled corticosteroid, Global Initiative on Chronic Obstructive Lung Disease stage, region, COPD Assessment Test score (replacing baseline symptom score), exacerbations treated with antibiotics/steroids history in previous year (replacing 1-year history of exacerbations); Test type: Superiority; p = 0.0010, Negative binomial model; Ratio of rates = 0.89, 95% CI 2-sided [0.84 to 0.96] — Ratio of rates Tiotropium (5 μg) versus Tiotropium (5 μg) + Olodaterol (5 μg) is provided
Statistical Analysis 3: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); Model was based on HERMES- Covariates: age, sex, smoking status, baseline Long-acting Beta-agonist/inhaled corticosteroid, region and percent predicted post-bronchodilator Forced Expiratory Volume in One Second; Test type: Superiority; p = 0.0080, Negative binomial model; Ratio of rates = 0.91, 95% CI 2-sided [0.85 to 0.98] — Ratio of rates Tiotropium (5 μg) versus Tiotropium (5 μg) + Olodaterol (5 μg) is provided
Statistical Analysis 4: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); Model was based on TRINITY/TRILOGY- Covariates: Treatment, region, severity of airflow limitation, and smoking status as effects, and exacerbations treated with antibiotics/steroids in previous year; Test type: Superiority; p = 0.0011, Negative binomial model; Ratio of rates = 0.89, 95% CI 2-sided [0.84 to 0.96] — Ratio of rates Tiotropium (5 μg) versus Tiotropium (5 μg) + Olodaterol (5 μg) is provided

2. Secondary Outcome: Number of Patients With at Least One Moderate to Severe COPD Exacerbation During the Actual Treatment Period.
Description: Key secondary endpoint: Number of patients with at least one moderate to severe COPD exacerbation during the actual treatment period per treatment. The actual treatment period was defined as the interval from first in-take of study medication until 1 day after last in-take of study medication. The median was not estimated due to less than 50% of patients having an event. Hence the number of patients with at least one moderate to severe COPD exacerbation is presented.
Time Frame: From first in-take of study medication until 1 day after last in-take of study medication, up to 361 days
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
Number analyzed (Participants) | 3941 | 3939
Number of patients | 1777 | 1746
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); A Cox's proportional hazard model was used to estimate the hazard ratio and the corresponding Confidence Interval. A log-rank test was used to obtain the p-value; Test type: Superiority — This hypothesis testing strategy ensures that the overall type I error is protected at 2-sided 0.01 level; p = 0.1188, Log Rank; Hazard Ratio (HR) = 0.95, 99% CI 2-sided [0.87 to 1.03] — Tiotropium (5 μg) + Olodaterol (5 μg) versus Tiotropium (5 μg)

3. Secondary Outcome: Annualised Rate of Exacerbations Leading to Hospitalisation During the Actual Treatment Period.
Description: Annualised rate of exacerbations leading to hospitalisation during the actual treatment period was calculated per treatment per patient-year. The actual treatment period was defined as the interval from first in-take of study medication until 1 day after last in-take of study medication.
Time Frame: From first in-take of study medication until 1 day after last in-take of study medication, up to 361 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Rate per patient-year
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
Number analyzed (Participants) | 3941 | 3939
Rate per patient-year | 0.20 [0.18 to 0.22] | 0.18 [0.16 to 0.20]
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); Annualised rate of exacerbations leading to hospitalization was analysed using a negative binomial model including the fixed, categorical effect of treatment as well as the logarithm of the treatment exposure as an offset; Test type: Superiority; p = 0.1265, Negative binomial model; Ratio of events vs. Tiotropium 5 μg = 0.89, 95% CI 2-sided [0.76 to 1.03] — Ratio of events Tiotropium (5 μg) + Olodaterol (5 μg) versus Tiotropium (5 μg) is provided

4. Secondary Outcome: Number of Patients With at Least One COPD Exacerbation Leading to Hospitalisation During the Actual Treatment Period.
Description: Number of patients with at least one COPD exacerbation leading to hospitalisation during the actual treatment period per treatment. The actual treatment period was defined as the interval from first in-take of study medication until 1 day after last in-take of study medication. The median was not estimated due to less than 50% of patients having an event. Hence the number of patients with at least one moderate to severe COPD exacerbation leading to hospitalisation is presented.
Time Frame: From first in-take of study medication until 1 day after last in-take of study medication, up to 361 days
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
Number analyzed (Participants) | 3941 | 3939
Number of patients | 469 | 450
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2773, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.82 to 1.06] — Tiotropium (5 μg) + Olodaterol (5 μg) versus Tiotropium (5 μg)

5. Secondary Outcome: Number of Patients With All-cause Mortality Occurring During the Actual Treatment Period.
Description: Number of patients with all-cause mortality occurring during the actual treatment period per treatment. The actual treatment period was defined as the interval from first in-take of study medication until 1 day after last in-take of study medication. The median was not estimated due to less than 50% of patients having an event. Hence the number of patients with all-cause mortality is presented.
Time Frame: From first in-take of study medication until 1 day after last in-take of study medication, up to 361 days
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
Number analyzed (Participants) | 3941 | 3939
Number of patients | 32 | 36
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium (5 μg) + Olodaterol (5 μg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7357, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.67 to 1.75] — Tiotropium (5 μg) + Olodaterol (5 μg) versus Tiotropium (5 μg)

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication until 21 days after last in-take of trial medication, up to 381 days
Description: Safety analyses were based on the treated set, which included all randomised patients who took at least 1 dose of trial medication during the randomised treatment period. Patients were only actively requested to report adverse events during the on-treatment period.
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium (5 μg) + Olodaterol (5 μg)
All-Cause Mortality (participants affected / at risk) | 98/3941 | 92/3939
Serious Adverse Events (participants affected / at risk) | 862/3941 | 810/3939
Other Adverse Events (participants affected / at risk) | 1786/3941 | 1770/3939
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 5 Microgram (μg) (N=3941) | Tiotropium (5 μg) + Olodaterol (5 μg) (N=3939)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Accelerated idioventricular rhythm (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 4 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 9 | 11
Angina pectoris (Cardiac disorders) | 8 | 4
Angina unstable (Cardiac disorders) | 14 | 6
Aortic valve disease mixed (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 2 | 1
Arrhythmia (Cardiac disorders) | 2 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 12 | 18
Atrial flutter (Cardiac disorders) | 4 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 8 | 8
Cardiac failure (Cardiac disorders) | 21 | 23
Cardiac failure acute (Cardiac disorders) | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 5 | 5
Cardiac failure congestive (Cardiac disorders) | 14 | 17
Cardio-respiratory arrest (Cardiac disorders) | 6 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 3 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 2
Cor pulmonale (Cardiac disorders) | 5 | 5
Cor pulmonale acute (Cardiac disorders) | 1 | 1
Cor pulmonale chronic (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 11 | 8
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 1
Microvascular coronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocardial haemorrhage (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 13 | 10
Myocardial ischaemia (Cardiac disorders) | 3 | 3
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 1
Right ventricular failure (Cardiac disorders) | 2 | 3
Sinoatrial block (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 4
Tachycardia (Cardiac disorders) | 3 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 3
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Myocardial bridging (Congenital, familial and genetic disorders) | 0 | 1
Porokeratosis (Congenital, familial and genetic disorders) | 1 | 0
Retinal anomaly congenital (Congenital, familial and genetic disorders) | 0 | 1
Syringomyelia (Congenital, familial and genetic disorders) | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Age-related macular degeneration (Eye disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 3
Cataract subcapsular (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Gaze palsy (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 3 | 2
Macular degeneration (Eye disorders) | 0 | 2
Macular fibrosis (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 2
Open angle glaucoma (Eye disorders) | 2 | 0
Retinal tear (Eye disorders) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 3
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 4
Intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Necrotising colitis (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Subileus (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 3 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 11 | 10
Death (General disorders) | 14 | 3
Hyperplasia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Medical device site haematoma (General disorders) | 0 | 1
Medical device site pain (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 6 | 2
Non-cardiac chest pain (General disorders) | 0 | 3
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Peripheral swelling (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 4
Sudden cardiac death (General disorders) | 0 | 2
Sudden death (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 2
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 4
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 3
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Botulism (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 4
Bronchitis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 3
Chronic sinusitis (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Colon gangrene (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 3 | 0
Empyema (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 4 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Giardiasis (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4
Infected skin ulcer (Infections and infestations) | 1 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 15 | 15
Infective glossitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 10 | 1
Intestinal gangrene (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 3 | 1
Lung infection (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Oral bacterial infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 144 | 132
Pneumonia bacterial (Infections and infestations) | 3 | 3
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 3
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 10 | 9
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 5 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Strongyloidiasis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 2 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 12 | 3
Urosepsis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 3
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 12 | 10
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 1 | 0
Occupational exposure to product (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 2
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Petroleum distillate poisoning (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2
Stress fracture (Injury, poisoning and procedural complications) | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 4
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood lactic acid increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Breath sounds absent (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
PCO2 increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte depletion (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Cartilage hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 6
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 10
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung infiltration malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 13
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mucoepidermoid carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penis carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 8
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acoustic neuritis (Nervous system disorders) | 1 | 0
Alcohol induced persisting dementia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Anterior interosseous syndrome (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 3 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 3 | 2
Cerebral ischaemia (Nervous system disorders) | 2 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 7 | 8
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 0 | 3
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 2
Facial neuralgia (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Hemianaesthesia (Nervous system disorders) | 0 | 1
Hemianopia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 2 | 3
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 4 | 5
Lacunar stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Mononeuropathy (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 3 | 5
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 4
Tremor (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Device breakage (Product Issues) | 0 | 1
Device lead damage (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 2 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Brief psychotic disorder with marked stressors (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 2 | 3
Disorientation (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 15
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1
Renal salt-wasting syndrome (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 3 | 1
Urethral fistula (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 4
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 4
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 | 21
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 405 | 394
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 43 | 33
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Enterostomy (Surgical and medical procedures) | 0 | 1
Gallbladder operation (Surgical and medical procedures) | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 1
Lung transplant (Surgical and medical procedures) | 0 | 1
Pancreatic operation (Surgical and medical procedures) | 0 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 3 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 3
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Brachiocephalic arteriosclerosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 3 | 3
Deep vein thrombosis (Vascular disorders) | 8 | 1
Embolism (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 5 | 3
Hypertensive crisis (Vascular disorders) | 9 | 6
Hypotension (Vascular disorders) | 2 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Macroangiopathy (Vascular disorders) | 0 | 1
Microscopic polyangiitis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 3
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 2
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 1 | 1
Subgaleal haematoma (Vascular disorders) | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 5 Microgram (μg) (N=3941) | Tiotropium (5 μg) + Olodaterol (5 μg) (N=3939)
Viral upper respiratory tract infection (Infections and infestations) | 293 | 281
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1504 | 1519
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 232 | 203

LIMITATIONS AND CAVEATS:
One site was closed for cause due to data irregularities. The data from the 21 patients at this site were excluded from the patient sets used for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02296138/SAP_000.pdf
  • Study Protocol (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02296138/Prot_001.pdf